CLINICAL TRIAL: NCT03263494
Title: CGM Intervention in Teens and Young Adults With T1D (CITY): A Randomized Clinical Trial to Assess the Efficacy and Safety of Continuous Glucose Monitoring in Young Adults 14-<25 With Type 1 Diabetes
Brief Title: CGM Intervention in Teens and Young Adults With Type 1 Diabetes (T1D)
Acronym: CITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CITY
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CGM (Active Comparator)
  Interventions: Device: Continuous Glucose Monitor (CGM)
- BGM (No Intervention)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — Participants randomized to the CGM Group will receive a Dexcom CGM device and be instructed on how to utilize the CGM data in real time for diabetes management.
  Arms: CGM

SUMMARY:
Adolescents and young adults with T1D and poor glycemic control (age 14-< 25 years, T1D duration >12 months, HbA1c 7.5-<11.0%, using an insulin pump or MDI)) will be randomly assigned to either CGM or BGM. Sample size will be 150. The primary outcome assessment will be HbA1c after 6 months. Secondary outcomes will include HbA1c, CGM metrics (control group will wear blinded CGM at 13 and 24 weeks), and quality of life measures. The randomized trial will be followed by a 6-month extension study during which the RCT control group will initiate CGM and the RCT CGM group will continue CGM.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of T1D, with either age of T1D diagnosis < 10 years of age OR a history of positive T1D related antibodies in the medical record
2. Age 14-<25 years
3. Diabetes duration ≥ 1 year
4. Total daily insulin requirement ≥ 0.4 units/kg/day
5. HbA1c 7.5% to <11.0% (Point of care device or local lab measured as part of study at screening visit)
6. Insulin regimen involves a consistent modality of insulin administration with either use of an insulin pump or at least 3 multiple daily injections of basal and bolus (meal time) analogue insulin. Insulin pump must not have been started within 3 months of consent with no plans to change regimens in the next 6 months
7. Perform at least 2 blood glucose meter checks per day from self-report at screening and an average of at least 2 checks per day from meter download during blinded CGM run in
8. Blinded CGM must be used a minimum of 200 hours (equivalent to 8.3 days) with an average of 1.8 calibrations per day during the blinded CGM screening period.
9. Participant comprehends written and spoken English
10. Participant understands the study protocol and agrees to it (if applicable)

Exclusion Criteria:

1. Use of unblinded personal CGM and/or flash CGM, outside of a research study, as part of real-time diabetes management in the last 3 months
2. Unable to use CGM device for minimum number of hours during blinded pre-randomization period or skin reaction from adhesive that would preclude participation in the randomized trial
3. Started on non-insulin medication for blood glucose control within the past 3 months or plans to begin within the next 6 months
4. The presence of a significant medical disorder that in the judgment of the investigator will affect the wearing of the sensors (such as a skin condition), or the completion of any aspect of the protocol.
5. More than 1 episode of DKA in the past 6 months as defined in the adverse events chapter.
6. The presence of any of the following diseases:

   * Asthma or any condition present in the last 6 months where treatment is a systemic or daily inhaled corticosteroid (Intermittent treatment with inhaled corticosteroids does not exclude subjects from enrollment)
   * Cystic fibrosis
   * Addison's disease (Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment)
7. Inpatient psychiatric treatment in the past 6 months or daily intensive outpatient psychiatric day treatment in the past 3 months.
8. Pregnant (positive test confirmed at screening) or planning to become pregnant in the next 12 months.
9. Need for use of acetaminophen or acetaminophen-containing products on a regular basis during the 6 months of the trial
10. Participation in a diabetes related intervention study in the past 6 weeks.
11. Any medical, psychological or social situation where per investigator discretion it may be difficult for participant to participate fully in the intervention
12. Any condition, per investigator assessment, that could impact reliability of the A1C measurement, such as (but not limited to) hemoglobinopathy, hemolytic anemia, chronic liver disease; chronic GI blood loss, red blood cell transfusion or erythropoietin administration within 3 months prior to screening

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to 26 weeks adjusted for baseline | 6 months

SECONDARY OUTCOMES:
% with HbA1c <7.0% | 6 months
% with HbA1c <7.5% | 6 months
% with relative reduction ≥ 10% | 6 months
% with absolute reduction ≥ 0.5% | 6 months
% with absolute reduction ≥ 1% | 6 months
% with absolute reduction ≥ 1% or HbA1c < 7.0% | 6 months
CGM % time in range 70-180 mg/dl | 6 months
CGM mean glucose | 6 months
CGM glucose variability measured by coefficient of variation | 6 months
CGM % time > 180 mg/dl | 6 months
CGM % time > 300 mg/dl | 6 months
CGM % time < 54 mg/dl | 6 months
CGM % time < 70 mg/dl | 6 months
Rate of CGM measured hypoglycemic episodes (using <54 mg/dL) | 6 months
CGM Self Efficacy Questionnaire Score | 6 months
  Questionnaire containing 15 questions with possible responses 0-6. Total score is calculated by taking the mean of the non-missing responses. Then multiply by 100 and divide by 6 to put on the scale 0-100. Higher total score indicates higher perceived ability.
Problem Areas in Diabetes (PAID) Questionnaire Score | 6 months
  Survey containing 20 questions with possible responses 0-5. Total score is calculated by taking the mean of the non-missing items and multiplying by 20 to put on the scale 0-100. A higher total score indicates more of a problem.
Glucose Monitoring Satisfaction Questionnaire Score | 6 months
  Survey containing 15 questions. Total score ranges from 0-100. A higher total score indicates more satisfaction with their current glucose monitor.
Hypoglycemia Confidence Questionnaire Score | 6 months
  Survey containing 9 questions with possible responses 0-4. Total score is calculated by taking the mean of non-missing responses and multiplying by 25 to put on the scale 0-100. Higher total score indicates more confidence.
Diabetes Technology Attitudes Questionnaire Score | 6 months
  Survey containing 5 questions with possible responses 0-4. Total score is calculated by taking the mean of non-missing responses and multiplying by 25 to put on the scale 0-100. Higher total score indicates a more positive attitude towards diabetes technology.
Pittsburgh Sleep Quality Index | 6 months
  Survey containing 19 questions. Total score ranges from 0-21. A lower score indicates a healthier sleep quality.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Barbara Davis Center--University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Joslin Diabetes Center, Boston, Massachusetts
  - IDC at Park Nicollet, Saint Louis Park, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Naomi Berrie Diabetes Center at Columbia University, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller KM, Bauza C, Kanapka LG, Clements MA, DeSalvo DJ, Hood K, Messer LH, Sherr J, Bergamo K, Criego A, Freiner E, Lyons SK, Monzavi R, Moore W, Prahalad P, Simmons JH, Sulik M, Wadwa RP, Weinstock RS, Willi SM, Williams K, Laffel LM; CITY Study Group. Continuous Glucose Monitoring Provides Durable Glycemic Benefit in Adolescents and Young Adults with Type 1 Diabetes: 12-Month Follow-Up Results. Pediatr Diabetes. 2023 Oct 26;2023:6718115. doi: 10.1155/2023/6718115. eCollection 2023. PMID 40303270
- [Derived] Laffel LM, Kanapka LG, Beck RW, Bergamo K, Clements MA, Criego A, DeSalvo DJ, Goland R, Hood K, Liljenquist D, Messer LH, Monzavi R, Mouse TJ, Prahalad P, Sherr J, Simmons JH, Wadwa RP, Weinstock RS, Willi SM, Miller KM; CGM Intervention in Teens and Young Adults with T1D (CITY) Study Group; CDE10. Effect of Continuous Glucose Monitoring on Glycemic Control in Adolescents and Young Adults With Type 1 Diabetes: A Randomized Clinical Trial. JAMA. 2020 Jun 16;323(23):2388-2396. doi: 10.1001/jama.2020.6940. PMID 32543683

DOCUMENTS (1):
  • Informed Consent Form (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT03263494/ICF_000.pdf